CLINICAL TRIAL: NCT05988788
Title: Effect of Epigallocatechin-3-Gallate Solution Versus Sodium Hypochlorite as a Root Canal Irrigant on Post-Operative Pain Intensity and Bacterial Load Reduction in Asymptomatic Necrotic Mandibular Premolars: A Randomized Clinical Trial
Brief Title: Effect of Epigallocatechin-3-Gallate Solution as a Root Canal Irrigant on Post-Operative Pain Intensity and Bacterial Load Reduction in Necrotic Tooth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rayan Elsadig Izzeldin, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Epigallocatechin-3-Gallate
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Necrotic Pulp
Keywords: Asymptomatic; Necrotic Mandibular premolar
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — epigallocatechin gallate; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Epigallocatechin-3-Gallate (Experimental): 20% Epigallocatechin-3-Gallate solution
  Interventions: Other: Epigallocatechin-3-gallate
- sodium hypochlorite (Active Comparator): 2.5% sodium hypochlorite
  Interventions: Other: sodium hypochlorite

INTERVENTIONS:
Other: Epigallocatechin-3-gallate — to be used as a root canal irrigant
  Other Names: green tea catechin
  Arms: Epigallocatechin-3-Gallate
Other: sodium hypochlorite — to be used as a root canal irrigant
  Arms: sodium hypochlorite

SUMMARY:
clinically compare the intensity of post-operative pain and the amount of bacterial load reduction after using 20% Epigallocatechin-3-gallate solution during chemomechanical preparation, versus 2.5% NaOCl, in asymptomatic necrotic mandibular premolars treated in a single visit.

DETAILED DESCRIPTION:
The patients will be randomly divided into 2 groups. Intervention group (20% epigallocatechin-3-gallate solution root canal irrigant) and control group (2.5% sodium hypochlorite root canal irrigant).

Post-operative pain will be measured at 6, 12, 24 and 48 hours post-operatively. The pain will be recorded using the Numerical Rating Scale (NRS).

Amount of bacterial load reduction The intracanal bacterial load reduction will be determined using agar culture technique by counting the colony forming units per milliliter (CFUs/mL) before and after root canal preparation.

ELIGIBILITY:
The inclusion criteria:

1. Systematically healthy patient (ASA I, II).
2. Age between 18 and 45 years
3. Male or female.
4. Asymptomatic mandibular premolar teeth diagnosed with pulp necrosis.

The exclusion criteria:

1. Medically compromised patients having significant systemic disorders. (ASA III or IV).
2. Teeth with:

   * Immature roots
   * Association with swelling or sinus tract.
   * Acute peri-apical abscess or acute exacerbation of a chronic abscess.
   * Mobility Grade II or III
   * Previously accessed or endodontically treated
   * Deep periodontal pockets more than 4 mm
   * Vertical root fractures, coronal perforation, calcification, and external or internal root resorptions.
3. Patients who could not interpret the NRS.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative pain measured at 6, 12, 24, 48 hours after single visit treatment.
  Categorical None 0 Mild 1-3 Moderate 4-6 Severe 7-10

SECONDARY OUTCOMES:
Amount of intracanal bacterial load reduction | T0: preintervention, preinstrumentation after access cavity. T1: postinstrumentation up to 10 min
  The intracanal bacterial load reduction will be determined using agar culture technique by counting the colony forming units per milliliter (CFUs/mL) before and after root canal preparation

CONTACTS AND LOCATIONS:
Overall Officials: rayan adlan, Principal Investigator — Cairo University
Locations (1):
- Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF